CLINICAL TRIAL: NCT07044128
Title: Prospective, Controlled, Open-label Study Evaluating the Keikku Electronic Stethoscope
Brief Title: Validate the Efficacy and the Safety of the Keikku Electronic Stethoscope for Its Indication and Intended Purpose, Under the Intended Conditions of Use.
Acronym: KCI-1
Status: Recruiting | Type: Observational
Sponsor: Lapsi Health Holding B.V. (Industry)
Collaborators: Clínica Internacional (Other)
Responsible Party: Sponsor
Other Study IDs: D087
Record Dates: First submitted 2025-06-23; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Heart Murmurs; Wheezing
Keywords: Stethoscopes; Heart Murmurs; Cardiac Auscultation; Diagnostic Techniques and Procedures; Medical Device Evaluation; Sound Recording and Reproduction; Pediatric Cardiology; Adult Cardiology; Telemedicine; Signal Processing, Computer-Assisted; Electronic Health Records; Clinical Accuracy; Safety Assessment; Prospective Studies
MeSH Terms: conditions — Heart Murmurs; Respiratory Sounds | interventions — Heart Auscultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Keikku Stethoscope Evaluation Group - Pediatric: This group includes pediatric participants undergoing non-urgent cardiac evaluation. Each participant receives heart sound assessments using both the investigational Keikku electronic stethoscope and a conventional analog stethoscope. The primary aim is to compare the accuracy of murmur detection between the two devices. Evaluations are performed by two separate physicians to ensure independent assessment.
  Interventions: Device: Digital stethoscope using MEMS sensor and mobile application for cardiac auscultation
- Keikku Stethoscope Evaluation Group - Adults: This group includes adult participants undergoing non-urgent cardiac evaluation. Each participant receives heart sound assessments using both the investigational Keikku electronic stethoscope and a conventional analog stethoscope. The primary aim is to compare the accuracy of murmur detection between the two devices. Evaluations are performed by two separate physicians to ensure independent assessment.
  Interventions: Device: Digital stethoscope using MEMS sensor and mobile application for cardiac auscultation

INTERVENTIONS:
Device: Digital stethoscope using MEMS sensor and mobile application for cardiac auscultation — The intervention is a digital stethoscope system comprising a handheld device with a micro-electromechanical system (MEMS) sensor and a Bluetooth Low Energy (BLE) connection to a mobile application (Keikku Mobile App) installed on an iOS or Android smartphone. The device captures auscultation sounds from standard precordial locations (mitral, tricuspid, aortic, and pulmonary), transmits them in real time to the mobile application, and stores the recordings on a secure, GDPR-compliant cloud server. The device does not interpret sounds. Each auscultation lasts 15 seconds per site. Physicians use Bluetooth headphones to listen during recording. The application allows for annotation and review of sound data. The intervention is administered once per participant during a single study visit, immediately followed by a comparator auscultation using a conventional analog stethoscope by a second blinded physician.

SUMMARY:
This study is testing a digital stethoscope called the Keikku electronic stethoscope. Doctors use stethoscopes to listen to the heart, and this new device records heart sounds using a smartphone app. The purpose of the study is to check how well this new device works and whether it is safe to use.

The study will include 149 participants of all ages (from birth to 99 years), who are undergoing routine (non-urgent) heart checks. After giving consent, each participant will have their heart sounds listened to twice: once with the Keikku electronic stethoscope and once with a regular stethoscope. Two different doctors will do the listening, and they won't share information with each other. The doctors will record whether they hear a heart murmur and how clear the sounds were.

The study will compare the findings from the new device to those from the regular stethoscope. Researchers will also check for any device problems or side effects. The study takes place at a single site in Peru and will take about one day for each participant.

The goal is to find out if the Keikku electronic stethoscope is accurate and safe for doctors to use in real medical settings.

DETAILED DESCRIPTION:
This clinical study is designed to evaluate the performance and safety of the Keikku electronic stethoscope, an innovative medical device developed by Lapsi Health Holding BV. The Keikku device combines a micro-electromechanical system (MEMS) sensor with a Bluetooth-enabled smartphone application, allowing physicians to capture and review heart sounds in real-time or via secure cloud storage.

The Keikku electronic stethoscope differs from traditional stethoscopes in that it digitally records and transmits auscultation sounds without interpreting them. Physicians use the Keikku Mobile Application to listen, annotate, and share these sounds. This study assesses whether such a device can match the diagnostic capabilities of conventional analog stethoscopes, particularly in detecting heart murmurs.

This is a prospective, open-label, controlled clinical investigation involving 149 pediatric and adult participants (from birth to age 99) in non-urgent cardiac evaluations. Each participant undergoes two sequential heart sound assessments at four standard precordial chest locations (mitral, tricuspid, aortic, and pulmonary):

Keikku electronic stethoscope: used by a physician listening via Bluetooth headphones.

Conventional stethoscope: used by a second, blinded physician.

Each device's use is independently evaluated using predefined clinical report forms. Physicians record whether a murmur is present and rate the acoustic quality of the auscultation on a 5-point Likert scale.

To ensure objectivity, physicians do not communicate their findings, and the second physician has no access to the recordings or results obtained by the first. All recordings (both digital and analog) are stored on GDPR-compliant cloud servers. Final clinical decisions about patient care are based only on the findings of the conventional stethoscope, not the investigational device.

The study's primary endpoint is the agreement percentage between the Keikku and conventional stethoscopes in murmur detection. Secondary and exploratory endpoints include the incidence of device-related adverse events, the sensitivity and specificity of murmur detection, user-reported sound quality, and any technical issues (device deficiencies) encountered.

Participation in this study lasts only one day and involves no follow-up visits. No treatment decisions are made based on the investigational device. The research is conducted at a single site in Peru, and the data will contribute to a broader understanding of digital stethoscope performance in clinical environments.

By validating the diagnostic capabilities of the Keikku electronic stethoscope, this study aims to support the safe integration of digital auscultation technology into everyday clinical care and remote telemedicine applications.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric, including newborn (from birth to 1 month of age), or adult (aged 99 or below) individuals.
* Individuals who are either:

  * presenting for initial, non-urgent outpatient evaluation of a cardiac murmur or for non-urgent cardiac clearance; or
  * presenting for return, non-urgent outpatient evaluation of a cardiac murmur; or
  * undergoing initial or recurrent, non-urgent evaluation of a cardiac murmur in inpatient setting; or
  * undergoing non-urgent cardiac clearance in inpatient setting.

Exclusion Criteria:

pregnant female individuals

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll 149 pediatric and adult male and non-pregnant female individuals, from birth to (and including) 99 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Agreement in murmur detection between digital and conventional stethoscopes | Day 0 (Single visit)
  Overall agreement (in percent) between the Keikku electronic stethoscope and a conventional analog stethoscope in identifying the presence or absence of a heart murmur.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Internacional San Borja, Lima, Peru

IPD SHARING:
Plan to Share IPD: No